CLINICAL TRIAL: NCT01744522
Title: Pilot Study on the Influence of Leech Therapy on Pain and Sensory Processing in Patients With Postherpetic Neuralgia
Brief Title: Leech Therapy for Postherpetic Neuralgia
Acronym: ZoHir
Status: Terminated | Type: Observational
Why Stopped: We were not able to recruit enough patients for this study within a given time frame.
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principal Investigator, Universität Duisburg-Essen
Other Study IDs: 12-5147-BO
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Leeching

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Leech therapy: Patients receiving leech therapy in the outpatient clinic
  Interventions: Procedure: Leech therapy

INTERVENTIONS:
Procedure: Leech therapy — Leech therapy: Using medicinal leeches After piercing the skin and injecting anticoagulants (hirudin) and anaesthetics, they suck out blood of the incision. After 30 to 60 minutes they fall off and the wound -after a short time of after-bleeding- is bandaged up.
  Other Names: Hirudo medicinalis; Leeching

SUMMARY:
The purpose of this study is to investigate, whether leech therapy for the treatment of postherpetic pain improves pain and sensory function.

Therefore 20 patients with PHN undergoing leech therapy at the investigators outpatient clinic will be included in this observational trial.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years of age
* >6 months thoracal postherpetic neuralgia
* informed consent

Exclusion Criteria:

* if leech therapy is contraindicated
* physical and mental disability to participate in the study examinations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from an outpatient clinic for naturopathy, traditional chinese and indian medicine(secondary care)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 28 days
  Pain intensity measured on a visual analogue scale (0-100mm, 100mm indicating worst pain imaginable)

SECONDARY OUTCOMES:
Pain intensity | 3 months
  pain intensity on a 100mm Visual Analogue Scale
Pain quality | 28 Days
  sensory and affective dimensions of pain (measured by the McGill Pain Questionnaire)
Pain quality | 3 months
  sensory and affective dimensions of pain (measured by the McGill Pain Questionnaire)
Impairment | 28 days
  functional impairment due to zoster pain, measured bey the zoster brief pain inventory and the zoster impact questionnaire (Coplan P, Schmader K, Nikas A, Chan I, Choo P, Levin M, Johnson G, Bauer M, Williams HM, Kapla KM, Guess HA, Oxman MN. (2004). Development of a measure of the burden of pain due to herpes zoster and postherpetic neuralgia for prevention trials: adaptation of the brief pain inventory. J Pain, 5(6), 344-356.)
Impairment | 3 months
  functional impairment due to zoster pain, measured bey the zoster brief pain inventory and the zoster impact questionnaire (Coplan P, Schmader K, Nikas A, Chan I, Choo P, Levin M, Johnson G, Bauer M, Williams HM, Kapla KM, Guess HA, Oxman MN. (2004). Development of a measure of the burden of pain due to herpes zoster and postherpetic neuralgia for prevention trials: adaptation of the brief pain inventory. J Pain, 5(6), 344-356.)
Quality of life | 28 days
  quality of life measured by the SF36
quality of life | 3 months
  quality of life measured by the SF36
Sensory perception and pain thresholds | 28 days
  Sensory perception and pain thresholds measured by the quantitative sensory testing battery (Rolke, R., Magerl, W., Campbell, K. A., Schalber, C., Caspari, S., Birklein, F. and Treede, R.-D. (2006), Quantitative sensory testing: a comprehensive protocol for clinical trials. European Journal of Pain, 10: 77.)
Sensory perception and pain thresholds | 3 months
  Sensory perception and pain thresholds measured by the quantitative sensory testing battery (Rolke, R., Magerl, W., Campbell, K. A., Schalber, C., Caspari, S., Birklein, F. and Treede, R.-D. (2006), Quantitative sensory testing: a comprehensive protocol for clinical trials. European Journal of Pain, 10: 77.)
Safety | 28 days
  all adverse and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Romy Lauche, PhD, Principal Investigator — Research fellow
Locations (1):
- Chair of Complementary and Integrative Medicine, Essen, Germany